CLINICAL TRIAL: NCT00785720
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd PH_DETINBACK (Lactic Acid) Sweet Flower
Brief Title: Dermacyd PH_DETINBACK (Lactic Acid) Sweet Flower - Photo Avaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04303
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Dermacyd PH_DETINBACK (Lactic Acid)
  Interventions: Drug: Dermacyd PH_DETINBACK (Lactic Acid)

INTERVENTIONS:
Drug: Dermacyd PH_DETINBACK (Lactic Acid)

SUMMARY:
The purpose of this study is to demonstrate the absence of photoirritation and photosensitization potential of the product Dermacyd PHDETINBACK Sweet Flower.

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin II and III;
* Integral skin test in the region;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs 15 days before the selection;
* Diseases which can cause immunity decrease, such as HIV, diabetes;
* Use of drug photosensitizer;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease which can change the study results;
* History of photodermatosis active;
* Family or personal antecedent of cutaneous photoinduced neoplasias;
* Presence of a precursor lesion of cutaneous neoplasia, such as nevus melanocyte and queratoses actinium;
* Intense solar exposure in the study area;
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The photo irritation test and the photosensitivity will be measured using UVA irradiation and evaluated according International Contact Dermatitis Research Group (ICDRG) scale. The sensibility will be evaluated according to the skin type. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil